CLINICAL TRIAL: NCT05444114
Title: What Makes People Better at Describing Photographs?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Colorado Springs (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lori James, Professor, University of Colorado, Colorado Springs
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020-006; R15AG063111-01 (NIH)
Record Dates: First submitted 2022-06-18; First posted 2022-07-05 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Healthy Aging
Keywords: speech production; cognitive aging

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two conditions before performing a picture description task from which we measure speech fluency in several ways
Who Masked: Participant
Masking Description: Participants in each condition do not know what other participants are doing, nor that there is another condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Breathing (Experimental): Participants follow instructions regarding a mindful breathing exercise on a 10-min audio clip
  Interventions: Behavioral: Mental Exercise
- Control (Active Comparator): Participants follow instructions and listen to a 10-min audio clip of a story
  Interventions: Behavioral: Mental Exercise

INTERVENTIONS:
Behavioral: Mental Exercise — Participants perform a 10 minute mental exercise that is either mindful breathing or listening to a story

SUMMARY:
This study is being conducted to learn more about how various personal and situational characteristics are related to the ability to provide verbal descriptions of photographs. Participants will perform a brief mental exercise, then see three photographs with instructions to describe each thoroughly. Participants will also complete several other surveys and measures. Collected data will give researchers a better understanding of how different variables relate to speech production.

DETAILED DESCRIPTION:
This study is being conducted to learn more about how various personal and situational characteristics are related to the the ability to provide verbal descriptions of photographs. Adult participants ages 18-30 and 65-80 will participate in videoconference calls during which they perform a brief mental exercise, then see three photographs with instructions to describe each thoroughly. Descriptions are to be 30 to 60 seconds in length and are audio recorded for later scoring. Participants will also complete several other surveys and measures, including some about anxiety, mindfulness, vocabulary, and demographics. Participation will take approximately 40 to 60 minutes. Collected data will be de-identified, and the aggregate data will give researchers a better understanding of how individuals' personality and cognitive traits and the mental exercise performed before the study relate to peoples' speech production performance.

ELIGIBILITY:
Inclusion Criteria:

* fluent speakers of English
* ages 18-30 or ages 65-80

Exclusion Criteria:

* non-fluent speakers of English
* people who are not ages 18-30 or ages 65-80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori James, PhD, Principal Investigator — University of Colorado, Colorado Springs
Locations (1):
- UCCS, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
De-identified participant data may be posted on a website for open access to other researchers, if the publication outlet requires it., but is not currently planned.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Young adult participants were recruited via an online posting system (Sona) operated within the UCCS Psychology department.
  Older adult participants were recruiting via calls and emails to community members who have signed up as interested in participating via a UCCS website.
Groups:
- Mindful Breathing Intervention: Participants followed along with a 10 minute mental exercise involving mindful breathing
- Control Condition: Participants listen to 10 minutes of a story told in relaxing style
Period: Overall Study
Arm/Group | Mindful Breathing Intervention | Control Condition
Started | 90 | 92
Analysis Population | 81 | 90
Completed | 90 | 92
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mindful Breathing Condition: Participants follow instructions on a 10-min audio clip
  Participants perform a 10 minute mindful breathing exercise
- Control Condition: Participants follow instructions on a 10-min audio clip
  Participants listen to 10 minutes of a story
- Total: Total of all reporting groups
Arm/Group | Mindful Breathing Condition | Control Condition | Total
Number analyzed (Participants) | 90 | 92 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 47 | 93
  >=65 years | 44 | 45 | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 63 | 129
  Male | 24 | 29 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 9 | 24
  Not Hispanic or Latino | 68 | 83 | 151
  Unknown or Not Reported | 7 | 0 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 3 | 13
  White | 69 | 78 | 147
  More than one race | 7 | 5 | 12
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Speech Rate
Description: Average number of words per second spoken
Time Frame: During the 40 to 60 minute experimental session
Population: 10 of the 182 tested participants' data were not analyzed (9 in mindful breathing and 1 in control condition) due to reporting ages outside our inclusion criterion (n = 2), reporting not being native English speakers (n = 3), excessive distraction during testing (n = 1), or equipment problems (n = 4).
Measure: Mean (Standard Deviation); unit: Words per Second
Groups:
- Mindful Breathing Condition: Participants performed a 10 minute mental exercise involving mindful breathing
- Control Condition: Participants listened to a peaceful 10 minute segment of a story
Arm/Group | Mindful Breathing Condition | Control Condition
Number analyzed (Participants) | 81 | 91
Words per Second | 2.12 (0.41) | 2.20 (0.35)

2. Primary Outcome: Speech Fillers Mid-Phrase
Description: Average number of mid-phrase speech fillers as a percentage of words spoken
Time Frame: During the 40 to 60 minute experimental session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of words spoken
Arm/Group | Mindful Breathing Condition | Control Condition
Number analyzed (Participants) | 81 | 91
percentage of words spoken | 1.5 (1.4) | 1.6 (1.5)

3. Primary Outcome: Speech Fillers Other
Description: Average number of speech fillers not in the middle of a phrase as a percentage of words spoken
Time Frame: During the 40 to 60 minute experimental session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of words with other fillers
Arm/Group | Mindful Breathing Condition | Control Condition
Number analyzed (Participants) | 81 | 91
percentage of words with other fillers | 4.4 (3.0) | 4.4 (2.1)

4. Primary Outcome: Repairs Plus False Starts
Description: Average number of repairs plus false starts as a percentage of words spoken. These two measures reflect the same underlying process so are summed together; indeed, one or the other term is sometimes used to indicate both measures.
Time Frame: During the 40 to 60 minute experimental session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of words with false starts
Arm/Group | Mindful Breathing Condition | Control Condition
Number analyzed (Participants) | 81 | 91
percentage of words with false starts | 1.3 (0.9) | 1.9 (1.1)

5. Primary Outcome: Repetitions
Description: Average number of repetitions as a percentage of words spoken
Time Frame: During the 40 to 60 minute experimental session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of words spoken with repeats
Arm/Group | Mindful Breathing Condition | Control Condition
Number analyzed (Participants) | 81 | 91
percentage of words spoken with repeats | 1.0 (0.9) | 1.4 (1.0)

ADVERSE EVENTS:
Time Frame: During the 1 hour experimental session
Description: This is a short, basic science, behavioral intervention with minimal risk.
Groups:
- Mindful Breathing: Participants performed a 10 minute mental exercise involving mindful breathing
- Control: Participants performed a 10 minute mental exercise in which they listened to a story
Arm/Group | Mindful Breathing | Control
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/92
Other Adverse Events (participants affected / at risk) | 0/90 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT05444114/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT05444114/SAP_001.pdf
  • Informed Consent Form (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT05444114/ICF_002.pdf